CLINICAL TRIAL: NCT01626963
Title: Randomised-controlled Trial on the Immune Response to Single-port Access Versus Conventional Laparoscopic Colorectal Surgery
Brief Title: Single-port Versus Conventional Laparoscopic Colorectal Surgery
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: North Tees and Hartlepool NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, David W Borowski, Consultant General and Colorectal Surgeon, North Tees and Hartlepool NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SUR-089
Record Dates: First submitted 2012-06-18; First posted 2012-06-25 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Colorectal Cancer; Inflammatory Bowel Disease; Benign Colorectal Neoplasm; Diverticular Disease
Keywords: single-port access; laparoscopic surgery; surgical trauma
MeSH Terms: conditions — Colorectal Neoplasms; Inflammatory Bowel Diseases; Diverticular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SPA (Experimental): Single-port access surgery
  Interventions: Procedure: Single-port access surgery
- CL (Active Comparator): Conventional Laparoscopic access
  Interventions: Procedure: Conventional Laparoscopic Access

INTERVENTIONS:
Procedure: Single-port access surgery — Surgery carried out through a single incision laparoscopic approach
  Arms: SPA
Procedure: Conventional Laparoscopic Access — Surgery through standard multiport laparoscopic approach
  Arms: CL

SUMMARY:
Conventional multi-port laparoscopic surgery (CL) is now a standard approach to colorectal resections, due to it's short-term benefits over conventional open surgery. In recent years, several studies have demonstrated that - in suitable patients - single-port access surgery (SPA) has similar clinical outcome compared to CL, with additional cosmetic benefits. It remains, however, unclear whether the trauma of surgery is also less for SPA compared to CL.

In this study, the investigators aim to randomise patients who are deemed suitable for SPA surgery to either SPA approach, or CL; in addition to clinical outcomes including length of operating time, post-operative pain scores, complications, quality of life indicators and cosmetic appearance, the investigators aim to compare the physiological response to trauma through biochemical markers (including C-reactive protein, White Blood Cell count) and cytokine expression (i.e. Interleukins IL-6 and IL-8). Patients will be analysed according to intention-to-treat analysis, with 25 patients in the SPA and 25 patients in the CL group. The patients will be operated by surgeons proficient in both CL and SPA surgery, and followed-up for the duration of their hospitalisation as well as at their routine out-patient visits, using questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* large bowel disorder requiring surgical resection
* body habitus suitable for single-port access surgery

Exclusion Criteria:

* patients not capable of informed consent and/or quality of life assessment
* planned open procedure for surgical reason
* multiple previous abdominal operations
* body-mass index > 40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-07 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Operative Time | assessment of electronic records at 30 days from surgery
  Operative Time

SECONDARY OUTCOMES:
Pain scores | change from baseline at 1,2,3,4 and 5 days from surgery
  Pain scores on visual Analog Scale
Complication / Conversion-to-open-surgery rates | assessment at 30 days post-op
  Complication / Conversion-to-open-surgery rates
Quality of Life indicators | change from baseline at 2, 4 weeks, & 3 months after surgery
  Quality of Life indicators
Cosmetic appearance | change from baseline at 2, 4 weeks and three months after surgery
  Body-Image scale
Cost comparison | assessment at the end of the study, up to 2 years post-op
  Assessment of overall cost, including theatre time, disposable equipment and length of hospital stay
LoS | assessment at 30 days from surgery
  Length of hospital stay
IL-6 | change from baseline at 2,6,24 and 72 hours from surgery
  Immune response to tissue trauma (Interleukin-6)
IL-8 | change from baseline at 2,6,24 and 72 hours from surgery
  Interleukin-8
WBCC | change from baseline at 2,6,24 and 72 hours from surgery
  White Blood Cell Count
CRP | change from baseline at 2,6,24 and 72 hours from surgery
  C-reactive Protein

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital North Tees, Stockton-on-Tees, United Kingdom